CLINICAL TRIAL: NCT01951053
Title: A Blinded, Placebo- and Comparator-Controlled Three-way Crossover Study to Investigate the Pharmacodynamics, Safety, Tolerability, and Pharmacokinetics of JNJ-40411813 in Healthy Male Subjects
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of JNJ-404118413 in Healthy Male Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: CR100064; 40411813EDI1003 (Other: Johnson & Johnson Pharmaceutical Research & Development); 2009-016637-95 (EudraCT Number)
Record Dates: First submitted 2013-08-27; First posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: Healthy; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; JNJ-40411813; Positive allosteric modulator
MeSH Terms: interventions — 1-butyl-3-chloro-4-(4-phenyl-1-piperidinyl)-(1H)-pyridone; Citalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Experimental): Participants will receive the study medications in the sequence of placebo, citalopram, and JNJ-40411813, in 3 treatment periods. Each treatment period has 3 days and subsequent treatment period will be separated by 7 days.
  Interventions: Drug: JNJ-40411813; Drug: Placebo; Drug: Citalopram
- Sequence 2 (Experimental): Participants will receive the study medications in the sequence of placebo, JNJ-40411813, and citalopram, in 3 treatment periods. Each treatment period has 3 days and subsequent treatment period will be separated by 7 days.
  Interventions: Drug: JNJ-40411813; Drug: Placebo; Drug: Citalopram
- Sequence 3 (Experimental): Participants will receive the study medications in the sequence of citalopram, placebo, and JNJ-40411813, in 3 treatment periods. Each treatment period has 3 days and subsequent treatment period will be separated by 7 days.
  Interventions: Drug: JNJ-40411813; Drug: Placebo; Drug: Citalopram
- Sequence 4 (Experimental): Participants will receive the study medications in the sequence of citalopram, JNJ-40411813, and placebo, in 3 treatment periods. Each treatment period has 3 days and subsequent treatment period will be separated by 7 days.
  Interventions: Drug: JNJ-40411813; Drug: Placebo; Drug: Citalopram
- Sequence 5 (Experimental): Participants will receive the study medications in the sequence of JNJ-40411813, placebo, and citalopram, in 3 treatment periods. Each treatment period has 3 days and subsequent treatment period will be separated by 7 days.
  Interventions: Drug: JNJ-40411813; Drug: Placebo; Drug: Citalopram
- Sequence 6 (Experimental): Participants will receive the study medications in the sequence of JNJ-40411813, citalopram, and placebo, in 3 treatment periods. Each treatment period has 3 days and subsequent treatment period will be separated by 7 days.
  Interventions: Drug: JNJ-40411813; Drug: Placebo; Drug: Citalopram

INTERVENTIONS:
Drug: JNJ-40411813 — Participants will receive nanosuspension of JNJ-40411813 500 mg orally once daily on Day 3 in appropriate treatment periods.
Drug: Placebo — Participants will receive placebo orally once daily on Days 1 to 2 or Days 1 to 3 in appropriate treatment periods.
Drug: Citalopram — Participants will receive citalopram 20 mg tablet orally once daily on Day 3 in appropriate treatment periods.

SUMMARY:
The purpose of the study is to evaluate the effect of JNJ-40411813 on rapid eye movement sleep and deep sleep; safety, tolerability and pharmacokinetics (what the body does to the study medication) of JNJ-40411813.

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor participants knows the treatment that the participant receives), placebo-controlled (effect of the study medication will be compared with the effect of placebo [inactive substance]), comparator-controlled (effect of the study medication will be compared with the effect of FDA approved and marketed active substance [citalopram]), and 3-way crossover (method used to switch participants from one treatment arm to another treatment arm) study. This study will be double-blinded for treatment with placebo and JNJ-40411813; however, it will be open label (all people know the identity of the intervention) for treatment with citalopram. This study will consist of screening phase (within 28 days prior to the start of study medication), treatment phase, and follow-up phase (approximately 14 days after the last administration of study medication). Participants will be randomly assigned to 1 of 6 sequences (Sequences 1, 2, 3, 4, 5, and 6) to receive JNJ-40411813, citalopram, and placebo. Each sequence consists of 3 treatment periods (Period 1, Period 2, and Period 3) and each subsequent treatment period will be separated by a wash out period (no treatment) of at least 7 days. Approximately, 18 participants will be enrolled in this study (3 participants in each sequence). Safety will be evaluated by the assessment of adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination which will be evaluated throughout the study duration. The total duration of study participation for a participant will be approximately 10 Weeks.

ELIGIBILITY:
Inclusion Criteria:

- Body mass index (BMI) between 18 and 29.9 kg/m2 (BMI is calculated as weight [kilogram] divided by square of height [meter])

Exclusion Criteria:

* Significant history of or current significant medical illness including (but not limited to) liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances or any other illness that the investigator considers clinically significant
* History of a relevant sleep disorder and / or receiving treatment for sleep disorders
* Regular or periodic use of benzodiazepines
* Serology positive for hepatitis B surface antigen, hepatitis C antibodies or HIV antibodies at screening
* Positive urine screen for drugs of abuse and positive alcohol breath test at screening or administration of the study medication
* Use of any prescription medication or over-the-counter medication (not including paracetamol), or herbal medication within 2 weeks of start of study medication

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Rapid Eye Movement (REM) sleep latency | Day 3 and Day 4
  REM sleep is a normal stage of sleep characterized by the rapid and random movement of the eyes. REM sleep latency is the time from sleep onset until first period of REM sleep. Polysomnographic recordings will be used to determine the time spent in different sleep stages (S1: light sleep, S2: light sleep, S3: deep sleep, and S4: REM sleep).
Total duration of Rapid Eye Movement (REM) sleep | Day 3 and Day 4
  Polysomnographic recordings will be used to determine the time spent in different sleep stages (S1: light sleep, S2: light sleep, S3: deep sleep, and S4: REM sleep). It will be calculated as number of epochs scored as REM sleep divided by 2.
Total time spent in deep sleep | Day 3 and Day 4
  Polysomnographic recordings will be used to determine the time spent in different sleep stages (S1: light sleep, S2: light sleep, S3: deep sleep, and S4: REM sleep). It will be calculated as number of stages score as 3 or stage 4 divided by 2.
Number of participants with adverse events as a measure of safety | Up to Week 10

SECONDARY OUTCOMES:
Peak plasma concentration of JNJ-40411813 | Day 3 (predose; 1, 3, 6, 14 and 16 hours post dose)
  This sample will be used for pharmacokinetics analysis.
Time to reach the peak plasma concentration of JNJ-40411813 | Day 3 (predose; 1, 3, 6, 14 and 16 hours post dose)
  This sample will be used for pharmacokinetics analysis.
Area under the plasma concentration of JNJ-40411813-time curve from 0 to t hours post dosing | Day 3 (predose; 1, 3, 6, 14 and 16 hours post dose)
  This sample will be used for pharmacokinetics analysis.
Area under the plasma concentration of JNJ-40411813-time curve from 0 to infinity post dosing | Day 3 (predose; 1, 3, 6, 14 and 16 hours post dose)
  This sample will be used for pharmacokinetics analysis.
Elimination rate constant of JNJ-40411813 | Day 3 (predose; 1, 3, 6, 14 and 16 hours post dose)
  This sample will be used for pharmacokinetics analysis.
Terminal half-life of JNJ-40411813 | Day 3 (predose; 1, 3, 6, 14 and 16 hours post dose)
  This sample will be used for pharmacokinetics analysis.
Time in bed | Day 3 and Day 4
  Time in bed is defined as time from 'lights out' to 'lights on'.
Latency to persistent sleep | Day 3 and Day 4
  Latency to persistent sleep is defined as time from 'lights out' to 'sleep onset'. Polysomnographic recordings will be used to determine the time spent in different sleep stages.
Sleep onset latency | Day 3 and Day 4
  Sleep onset latency is defined as time from 'lights out' to the beginning of 20 seconds epochs which have to be scored as sleep. Polysomnographic recordings will be used to determine the time spent in different sleep stages.
Total sleep time | Day 3 and Day 4
  Total sleep time is the duration of Rapid Eye Movement (REM) sleep plus non-REM sleep (sleep stages: S1: light sleep, S2: light sleep, and S3: deep sleep).
Sleep efficiency | Day 3 and Day 4
  Sleep efficiency is calculated as total sleep time divided by time in bed.
Number of awakenings | Day 3 and Day 4
  Number of awakenings is defined as number of stage shift from any sleep stage to wake. Polysomnographic recordings will be used to determine the time spent in different sleep stages.
Time spent awake after sleep onset | Day 3 and Day 4
  Time spent awake after sleep onset is defined as number of epochs scored as 'wake' (from the beginning of latency to persistent sleep until 'lights on'). Polysomnographic recordings will be used to determine the time spent in different sleep stages.
Duration of REM Sleep | Day 3 and Day 4
  Polysomnographic recordings will be used to determine the time spent in different sleep stages (S1: light sleep, S2: light sleep, S3: deep sleep, and S4: REM sleep).
Duration of Stage 1 Sleep | Day 3 and Day 4
  Duration of Stage 1 Sleep is the number of minutes spent in stage 1 from 'lights out' to 'lights on'. Polysomnographic recordings will be used to determine the time spent in different sleep stages.
Duration of Stage 2 Sleep | Day 3 and Day 4
  Duration of Stage 2 Sleep is the number of minutes spent in stage 2 from 'lights out' to 'lights on'. Polysomnographic recordings will be used to determine the time spent in different sleep stages.
Number of REM blocs | Day 3 and Day 4
  Number of REM blocs is defined as number of rapid eye movement episodes with a duration of at least 5 minutes. Polysomnographic recordings will be used to determine the time spent in different sleep stages (S1: light sleep, S2: light sleep, S3: deep sleep, and S4: REM sleep).

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Berlin, Germany